CLINICAL TRIAL: NCT03872245
Title: Association of Probiotics Intake With Percutaneous Electrical Neurostimulation of Dermatome T6 (PENS T6): Effect on Weight Loss in Obese Patients
Brief Title: Association of Probiotics With Neurostimulation of Dermatome T6: Effect on Weight Loss in Obese Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Garcilaso 19-3
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENS T6 + Probiotics (Experimental): The patients will receive Probiotics (Adomelle 1caps/12h) associated to PENS T6 during 10 weeks.
  Interventions: Biological: Probiotics; Procedure: PENS T6
- PENS T6 (Active Comparator): The patients will undergo PENS T6 during 10 weeks.
  Interventions: Procedure: PENS T6

INTERVENTIONS:
Biological: Probiotics — The patients will receive Adomelle 1caps/12h during 10 weeks
  Arms: PENS T6 + Probiotics
Procedure: PENS T6 — The patients will undergo percutaneous electrical neurostimulation of dermatome T6 weekle, during 10 weeks

SUMMARY:
Patients will be randomized into 2 groups:

* Group 1:Patients undergoing PENS T6, who also received Probiotics, during 10 weeks.
* Group 2: Patients undergoing PENS T6 during 10 weeks. They will not received Probiotics

Weight loss after 10 weeks of treatmente will be assessed.

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

* Group 1:Patients undergoing percutaneous electrical stimulation of dermatome T6 (PENS T6), who also received Probiotics (Adomelle 1 caps/12h), during 10 weeks.
* Group 2: Patients undergoing PENS T6 during 10 weeks. They will not received Probiotics

Weight loss after 10 weeks of treatmente will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 Kg/m2

Exclusion Criteria:

* Patients with pacemakers or implanted electrical devices.
* Pregnant women
* History of allergy to Probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-11 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 10 weeks
  Weight loss after treatment will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Llavero, Study Director — Hospital Rey Juan Carlos